CLINICAL TRIAL: NCT06725875
Title: Effects of White Noise and Earplugs Applied During Coronary Angiography on Patients' Physiological Parameters, Pain, Comfort and Procedure Satisfaction: A Randomized Controlled Experimental Study
Brief Title: Effects of White Noise and Earplugs on Patients' Physiological Parameters, Pain, Comfort and Procedure Satisfaction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Di̇lek Soylu (Other)
Responsible Party: Sponsor-Investigator, Di̇lek Soylu, Assistant professor, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/6674
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Coronary Angiography (CAG)
Keywords: White noise, earplug, coronary angiography, nurse, pain, comfort
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: White Noise Group — During the procedure, a mobile white noise (WN) application called Noise: White, Pink, Brown will be played via over-the-ear headphones to provide the individual with a sense of comfort. The intensity of the white noise will be determined using sound samples for patient comfort. The mobile WN application will be played to the patient by selecting white from among the color options. The sound level will be adjusted below 50 dB using a measuring device to prevent possible hearing damage (12). At the end of the procedure, the listening process will be terminated and the headphones will be removed. At the end of the procedure, the outer and inner surfaces of the headphones will be cleaned with disposable disinfectant wipes to prevent decontamination when used by another patient.
Other: Earplug group — 2. Earplug group: An earplug that prevents patients from hearing outside sounds will be used during the procedure. Features: Smooth, dirt-resistant surface provides better hygiene. Earplugs are easy to roll for quick and easy insertion. Conical design fits comfortably in ear canals. Soft polyurethane foam is hypoallergenic. Similar earplugs were used in a previous study

SUMMARY:
Coronary artery disease (CAD) is the leading cause of mortality and morbidity worldwide. Coronary Angiography (CAG) is an invasive method used in the diagnosis and treatment of CAD. Invasive methods such as coronary angiography cause pain. The sympathetic nervous system is stimulated and vital functions can be affected by the increased stress level of the pain experienced. In the angiography laboratory, patients are awake, aware of everything, and can easily hear the sounds of the monitor and the comments and conversations of the healthcare team. This auditory exposure can further trigger the patient's fear and anxiety and increase their pain. Increased anxiety can lead to an increase in the intensity of perceived pain and a decrease in pain tolerance. In addition to anxiety, catastrophizing such as fear of death can also be a means for disability and complications. In the literature, it is recommended to use nonpharmacological methods together with pharmacological treatment to increase pain tolerance and improve patient comfort and satisfaction in patients affected by invasive procedures. Nonpharmacological methods, unlike pharmacological agents, do not cause any harm to patients. It can help to keep physiological parameters such as blood pressure, respiration and pulse rate at normal levels and to increase comfort and satisfaction with the procedure. Sound therapy, which is a non-pharmacological method, turns the person's attention from negative stimuli to positive and hopeful feelings and can reduce stress, anxiety and pain.

Non-pharmacological methods such as white noise therapy and using earplugs that prevent sound permeability can be used to distract the patient's attention from the source of stress and focus on other thoughts. It is suggested that patients exposed to 50 to 55 dB white noise experience pain relief and have an effect on heart rate and oxygen saturation (12). As a result of our literature review, no studies were found where white noise was applied during coronary angiography. This situation reveals the originality of our study. With white noise, the patient can be isolated from ambient sounds during the procedure and the stress experienced can be controlled, the increase in pain intensity and decrease in tolerance that may occur due to stress can be controlled, and the patient's comfort and satisfaction level during the procedure can be increased. We think that the patient's compliance during the procedure can be increased.

The noise in the units affects the anxiety levels of the patients. The literature supports that the use of earplugs increases the comfort of the patient. In the study investigating the effect of auditory interventions on pain and comfort, it was determined that the pain level and heart rate were lower and the comfort level was higher in patients using earplugs compared to the control group. More evidence is needed on the effect of earplugs on physiological parameters, pain, comfort and procedure satisfaction of the patients by applying them to different patient groups. As a result of our literature review, no study was found where earplugs were applied during the coronary angiography procedure. This situation reveals another originality of our study.

The nurse involved in every step of coronary angiography aims to ensure that the patient benefits from the procedure to a high extent and to increase the quality of the procedure by integrating innovative methods. Nursing practices that increase the quality of the procedure are included in national and international nursing care guidelines. Therefore, in order to implement quality nursing care, it is necessary to increase the number of randomized controlled experimental studies and to increase the level of evidence. The fact that our study was a pre-test post-test randomized controlled double-blind study will increase the level of evidence in this regard. This situation reveals another originality of our study.

This study will use a randomized pre-test and post-test control group experimental design. It is planned that a total of 150 patients will participate in the study; 50 in the white noise group, 50 in the earplug group, and 50 in the control group. Data of the study will be collected via ''Personal information form, Numeric Pain Scale (NPS), Numeric Satisfaction Scale (NMS), Numeric Comfort Scale (NKS)''. A web-based randomization system will be used to determine the groups in the study. Pulse rate, respiratory rate, systolic blood pressure (SBP), diastolic blood pressure (DBP) and oxygen saturation values (SpO2) will be evaluated before, during, and after the procedure. Pain, satisfaction, and comfort levels will be evaluated at the end of the procedure. Interventions will be performed by the researcher and the patients will be observed throughout the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients who do not have vision, hearing, speech or comprehension problems, are 18 years of age or older, are open to communication and cooperation, do not have a psychiatric disease and agree to participate in the study will be included in the study.

Exclusion Criteria:

* Those with cognitive impairment or any auditory problems that may affect the test results, or those using psychoactive drugs will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2025-02-25 (Estimated); Study Completion 2025-02-25 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Scale | Immediate after angiography procedure
  The Numerical Pain Scale (NPS) was developed by Page et al (2012) (18) and will be used in this study to assess pain. The scale is a scale where the distance between two extreme points, with a minimum value of 0 at one end and a maximum value of 10 at the other end, is measured with a 10 cm ruler. In this context, the patient is explained that there are two extreme points and that he/she is free to mark any place between these points that is appropriate for the severity of his/her pain (5). The most important advantage of the test is that it does not have a language and is easy to apply. The horizontal or vertical line or length of the line on which the test is applied does not affect the measurement result. It is stated that the NAS is more sensitive and reliable than other single-dimensional scales in measuring pain intensity (19). Scala has been used in many studies (20), (5), (21).
Numerical Satisfaction Scale | Immediate after angiography procedure
  Patient satisfaction will be assessed using a numerical rating scale ranging from 0 to 10 points (0 = complete dissatisfaction, 10 = complete satisfaction). Previously used studies
Numerical Comfort Scale | Immediate after angiography procedure
  The comfort level of the patients will be evaluated using the (Numerical Rating Scale). In a previous validity and reliability study of the comfort scale (19), a similar scale validity was performed using the NRS while the validity and reliability study of the comfort scale was conducted and it was determined that the NRS could be used to evaluate the comfort level (21). In addition, other studies have evaluated the comfort level of the patients with the NRS. Patient comfort will be evaluated with a numerical rating scale between 0 and 10 points (0 = complete discomfort and 10 = complete comfort) (5), (21).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gokturk G, Sarialioglu A. Effect of white noise during nasal continuous positive airway pressure application on newborn's pain and stress levels, physiological parameters, and crying durations: A randomized controlled study. J Pediatr Nurs. 2024 Sep-Oct;78:e330-e337. doi: 10.1016/j.pedn.2024.07.022. Epub 2024 Jul 26. PMID 39060170
- [Background] Chaudhary A, Kumari V, Neetu N. Sleep Promotion among Critically Ill Patients: Earplugs/Eye Mask versus Ocean Sound-A Randomized Controlled Trial Study. Crit Care Res Pract. 2020 Dec 23;2020:8898172. doi: 10.1155/2020/8898172. eCollection 2020. PMID 33425385
- [Background] Bauersachs R, Zeymer U, Briere JB, Marre C, Bowrin K, Huelsebeck M. Burden of Coronary Artery Disease and Peripheral Artery Disease: A Literature Review. Cardiovasc Ther. 2019 Nov 26;2019:8295054. doi: 10.1155/2019/8295054. eCollection 2019. PMID 32099582